CLINICAL TRIAL: NCT03177993
Title: Community Based Safety Study of 2-drug (Diethylcarbamazine and Albendazole) Versus 3-drug (Ivermectin, Diethylcarbamazine and Albendazole) Therapy for Lymphatic Filariasis, Scabies and Soil Transmitted Helminths in Fiji
Brief Title: Fiji Integrated Therapy (FIT) - Triple Therapy for Lymphatic Filariasis, Scabies and Soil Transmitted Helminths in Fiji
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Task Force for Global Health (Other); Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201607068-2
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Lymphatic Filariases; Scabies; Impetigo; Soil Transmitted Helminths
MeSH Terms: conditions — Elephantiasis, Filarial; Scabies; Impetigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IDA 1 (Experimental): * ivermectin, diethylcarbamazine and albendazole Day 0,
  * permethrin Day 0 if excluded from ivermectin
  Details of dosing:
  * ivermectin: 200 mcg/kg oral
  * diethylcarbazine: 6mg/kg oral
  * albendazole 400mg oral
  * permethrin 5% cream topical: apply to whole body and wash o after 4hrs when less than 2 months; apply to whole body and wash off after 8hrs when 2 months and older.
  Interventions: Drug: 3 drug dose - IDA
- IDA 2 (Experimental): * ivermectin, diethylcarbamazine and albendazole Day 0, ivermectin Day 8
  * permethrin Day 0 and Day 8 if excluded from ivermectin
  Details of dosing:
  * ivermectin: 200 mcg/kg oral
  * diethylcarbazine: 6mg/kg oral
  * albendazole 400mg oral
  * permethrin 5% cream topical: apply to whole body and wash o after 4hrs when less than 2 months; apply to whole body and wash off after 8hrs when 2 months and older.
  Interventions: Drug: 3 drug dose - IDA with second dose of ivermectin
- DA (Active Comparator): * diethylcarbamazine and albendazole Day 0
  * permethrin Day 8 if scabies present in participant or household member
  Details of dosing:
  * diethylcarbazine: 6mg/kg oral
  * albendazole 400mg oral
  * permethrin 5% cream topical: apply to whole body and wash off after 4hrs when less than 2 months; apply to whole body and wash o after 8hrs when 2 months and older.
  Interventions: Drug: 2 drug dose - DA

INTERVENTIONS:
Drug: 3 drug dose - IDA — Lymphatic Filariasis Mass Drug Administration (MDA) with triple drug therapy of ivermectin, diethylcarbamazine, and albendazole (IDA). Participants excluded from ivermectin will receive a topical dose of permethrin cream.
  Exclusion criteria for ivermectin, diethylcarbamazine and albendazole:
  * severe illness (chronic renal insufficiency, severe chronic liver disease, or any illness that is severe enough to interfere with activities of daily living);
  * allergy to ivermectin, diethylcarbamazine or albendazole;
  * pregnant;
  * breastfeeding within 7 days of delivery;
  * less than 2 years old; OR
  * less than 15 kg
  In addition if less than 5 years old excluded from ivermectin.
  Exclusion criteria for permethrin:
  * allergy to permethrin
  * crusted scabies
  Other Names: IDA
  Arms: IDA 1
Drug: 3 drug dose - IDA with second dose of ivermectin — Lymphatic Filariasis Mass Drug Administration (MDA) with triple drug therapy of ivermectin, diethylcarbamazine, and albendazole (IDA). Eight days after treatment participants will be given a second dose of ivermectin alone.
  Participants excluded from ivermectin will receive a topical dose of permethrin cream both on day 0 and day 8.
  Exclusion criteria for ivermectin, diethylcarbamazine and albendazole:
  * severe illness (chronic renal insufficiency, severe chronic liver disease, or any illness that is severe enough to interfere with activities of daily living);
  * allergy to ivermectin, diethylcarbamazine or albendazole;
  * pregnant;
  * breastfeeding within 7 days of delivery;
  * less than 2 years old; OR
  * less than 15 kg
  In addition if less than 5 years old excluded from ivermectin.
  Exclusion criteria for permethrin:
  * allergy to permethrin
  * crusted scabies
  Other Names: IDA with second dose of ivermectin
  Arms: IDA 2
Drug: 2 drug dose - DA — Lymphatic Filariasis Mass Drug Administration (MDA) with the currently used standard of care combination drug therapy of diethylcarbamazine, and albendazole (DA).
  If scabies is present in the participant or a household member permethrin cream will be provided 8 days after dose of DA.
  Exclusion criteria for diethylcarbamazine and albendazole:
  * severe illness (chronic renal insufficiency, severe chronic liver disease, or any illness that is severe enough to interfere with activities of daily living);
  * allergy to diethylcarbamazine or albendazole;
  * pregnant;
  * breastfeeding within 7 days of delivery;
  * less than 2 years old; OR
  * less than 15 kg
  Exclusion criteria for permethrin:
  * allergy to permethrin
  * crusted scabies
  Other Names: DA
  Arms: DA

SUMMARY:
Lymphatic Filariasis (LF), scabies and soil transmitted helminths (STH) are common neglected tropical diseases affecting the people of Fiji. There is a dedicated LF eradication program supported by the World Health Organization (WHO), however scabies and STH are currently managed on an individual level with symptomatic treatment as required.

In an attempt to reduce the prevalence of LF globally, research is being undertaken into alternative, more effective treatment options. A recent study in Papua New Guinea demonstrated a new triple drug therapy (ivermectin, diethylcarbamazine and albendazole) is superior to the currently recommended two drug therapy (diethylcarbamazine and albendazole) used by WHO LF programs in the Pacific. However, adverse events were more frequent. Despite no serious adverse events being observed, it is necessary to conduct further studies to review the safety of this new triple therapy before it can be endorsed as an effective mass drug administration (MDA) regimen for LF in endemic countries. Fiji's burden of LF, that has been recalcitrant to previous MDA with diethylcarbamazine and albendazole, make it an ideal site to obtain further efficacy and safety data of the triple therapy.

Ivermectin given to communities as MDA has been proven to be effective in reducing the community prevalence of scabies. What is not known is the effects of one dose versus two doses of ivermectin as MDA. This question will be reviewed within the design of the community randomized study. The prevalence of impetigo in a community is linked to scabies and this will also be reviewed. Ivermectin and albendazole are both effective individually against STH. The effectiveness of this combination of treatment as MDA in Fiji for STH has not been studied. The effectiveness for the individual in the short-term and the community in the longer-term will be reviewed.

In addition, the acceptability and feasibility of the new therapy in communities at risk of these three diseases will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* All community members that have given written informed consent to participate

Exclusion Criteria:

* No informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4773 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Frequency, type, and severity of adverse events reported by participants following treatment with triple drug therapy (IDA) and standard two drug therapy (DA) in LF infected and uninfected individuals in a community as measured by CTCAE v4.03 | within 7 days of drug administration
  Participants will be interviewed and asked to report their general health status at baseline before receiving treatment and daily for the 2 days following treatment (Active Adverse Event Monitoring phase). For 3 to 7 days following treatment, anyone unwell the preceding day will be actively followed, other participants will be interviewed only if they feel unwell and present to the study team (Passive Adverse Event Monitoring phase).
  At any stage if they describe being unwell, further questions to determine type and severity of symptom(s) experienced will be asked and recorded according to pre-defined adverse event table. If participants report moderate to severe symptoms they will have further medical assessments as required.
  LF infection status will be determined by Filiarial Test Strip (FTS) and microfilariae (mf) smears.

SECONDARY OUTCOMES:
Clearance of microfilariae (mf) and filarial antigenemia following treatment with IDA or DA in LF infected individuals as measured by microfilaria count in 60ul thick blood smears and filarial test strip rapid diagnostic antigen test. | Baseline and 12 months
  Methods of assessment: FTS and Dried Blood Spot (DBS) for filarial antigenemia, mf smears for microfilariae
Prevalence of scabies in study population measured at baseline and 12 months after treatment using the WHO Integrated Management of Childhood Illness (IMCI) skin algorithm | Baseline and 12 months
  Methods of assessment: Skin examination
Prevalence of STH (hookworm, ascaris, trichuris and strongyloides) as measured by Kato-katz or PCR at baseline and 12 months after treatment | Stool collected at baseline (pre-treatment), 4 weeks (individual response), and 12 months (community prevalence).
  Methods of assessment: Stool samples will be analysed using Kato-katz method, as well as PCR.
Acceptability and feasibility of IDA and DA in communities at risk of LF, scabies and STH as assessed by survey and focus group discussions. | Approximately 4 weeks following treatment
  Methods of assessment: Acceptability Survey, designed specifically for the Triple therapy studies, Focus group discussions, Interviews with key informants
Prevalence of impetigo measured at baseline and 12 months after treatment using the WHO Integrated Management of Childhood Illness (IMCI) skin algorithm | Baseline and 12 months
  Methods of assessment: Skin examination

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Steer, PhD, Principal Investigator — Murdoch Childrens Research Institute; Gary Weil, MD, Principal Investigator — Washington University School of Medicine; Christopher King, MD PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Ministry of Health and Medical Services, Suva, Fiji

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publicly through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared publicly.

REFERENCES:
- [Derived] Hardy M, Samuela J, Kama M, Tuicakau M, Romani L, Whitfeld MJ, King CL, Weil GJ, Schuster T, Grobler AC, Engelman D, Robinson LJ, Kaldor JM, Steer AC. Community control strategies for scabies: A cluster randomised noninferiority trial. PLoS Med. 2021 Nov 10;18(11):e1003849. doi: 10.1371/journal.pmed.1003849. eCollection 2021 Nov. PMID 34758017
- [Derived] Hardy M, Samuela J, Kama M, Tuicakau M, Romani L, Whitfeld MJ, King CL, Weil GJ, Grobler AC, Robinson LJ, Kaldor JM, Steer AC. Individual Efficacy and Community Impact of Ivermectin, Diethylcarbamazine, and Albendazole Mass Drug Administration for Lymphatic Filariasis Control in Fiji: A Cluster Randomized Trial. Clin Infect Dis. 2021 Sep 15;73(6):994-1002. doi: 10.1093/cid/ciab202. PMID 33728462